CLINICAL TRIAL: NCT05497934
Title: The Effects of Glycerol as an Optical Clearing Agent for Visualization of the Middle Ear
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No response from initial letter or expiry email- closed by REB office
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Dalhousie University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1028201
Record Dates: First submitted 2022-08-10; First posted 2022-08-11 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Tympanosclerosis; Thickened Ears; Healthy; Surgery
MeSH Terms: conditions — Tympanosclerosis | interventions — Glycerol

STUDY DESIGN:
Intervention Model Description: All subjects will undergo OCT and conventional endoscopic imaging before topical application of glycerol to the tympanic membrane, after topical application of glycerol to the tympanic membrane and after rinsing the tympanic membrane with saline.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment arm (Experimental): Subjects will be imaged with OCT and endoscopy before treatment of the tympanic membrane with topical glycerol, after treatment of the tympanic membrane with topical glycerol and after rinsing the tympanic membrane with saline
  Interventions: Drug: Glycerol

INTERVENTIONS:
Drug: Glycerol — In this study, 99.5% pure glycerol will be used as an optical clearing agent. The glycerol will be applied topically to the tympanic membrane.
  Other Names: Glycerin(e)

SUMMARY:
This study will examine the improvement in middle ear optical coherence tomography imaging from the topical application of glycerol to the tympanic membrane in normal, opaque and post-operative ears

DETAILED DESCRIPTION:
This study will explore whether the utility of Optical Coherence Tomography (OCT) in otology patients can be enhanced through the application of topical glycerol as an optical clearing agent in patients with normal, opaque and post operative tympanic membranes. In each group of subjects, a comparison will be made between OCT images obtained before and after the topical application of glycerol to the tympanic membrane and following washout with saline. Images will also be assessed for their diagnostic utility as determined by the visibility of key structures and the change in middle ear mobility caused by glycerol absorption in the tympanic membrane.

ELIGIBILITY:
Inclusion Criteria:

* Thickened tympanic membrane (e.g. due to fibrosis) x10
* Tympanosclerosis of the tympanic membrane x10
* History of middle ear surgery with partial or total ossicular replacement prosthesis and cartilage tympanoplasty x10
* History of cartilage tympanoplasty without prosthesis implantation x10
* Normal tympanic membrane without history of middle ear disease x10

Exclusion Criteria:

* Narrow or stenotic external auditory canal that prevents visualization of the tympanic membrane
* Mobility disorder that prevents patient from remaining still during imaging
* Perforation of the tympanic membrane
* Open sores or infections of the external auditory canal

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in optical attenuation rate of the tympanic membrane | 20 minutes
  Change in optical attenuation rate (dB/mm) of the tympanic membrane between the pre-treatment and post-treatment conditions

SECONDARY OUTCOMES:
Change in acoustic mobility of the umbo | 20 minutes
  Change in the mobility (mm/s/Pa) of the umbo between pre- and post-treatment conditions
Change in B-mode signal-to-noise ratio of the cochlear promontorium | 20 minutes
  Change in the B-mode signal-to-noise ratio for a region of interest on the cochlear promontorium distal to the tympanic membrane between pre- and post-treatment conditions

CONTACTS AND LOCATIONS:
Overall Officials: David P Morris, MD, Principal Investigator — Nova Scotia Health Authority

IPD SHARING:
Plan to Share IPD: No
Results of trial will be published in a journal article